CLINICAL TRIAL: NCT06356753
Title: Association Between Chemical Exposome, Endometriosis and Infertility by an Integrative Approach
Brief Title: EndoxOmics : Exposome, Endometriosis and Fertility
Acronym: EndoxOmics
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0203
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis; Infertility, Female
Keywords: Exposome; Endometriosis; Infertility
MeSH Terms: conditions — Endometriosis; Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1-Women without deep endometriosis benefiting surgery: Group recruited from the gynaecology/obstetrics department : Women without deep endometriosis benefiting surgery.
  * Caucasian women, aged 18 to 45 years undergoing gynaecological surgery, for example: benign laparoscopy (example: tubal ligation), benign ovarian surgeries or benign uterine procedures (fibroma, ovarian cyst) or genital prolapse.
  * Non-interventional access to parietal and epiploic adipose tissue as part of routine care
  * No clinical-biological criteria in favour of a diagnosis of endometriotic disease, nor any radiological evidence (ultrasound or MRI) suggestive of endometriosis.
- 2-Women with endometriosis benefiting surgery: Group recruited from the gynaecology/obstetrics department : Women with endometriosis benefiting surgery.
  * Caucasian women aged 18 to 45
  * Severe and deep endometriotic pathology, with or without endometriomas, with surgical indication (clinical examination, imaging examinations, intraoperative observation),
  * Access to epiploid and/or parietal adipose tissue as part of routine care.
- 3-Infertile Women with deep endometriosis benefiting from IVF: Group recruited from the Reproductive Medicine Department : Infertile Women with deep endometriosis benefiting from IVF.
  * Women with IVF or ICSI for infertility with deep endometriosis diagnosed in routine care (clinical examination, imaging examinations +/- surgical findings). They will be classified into 2 subgroups: 1) deep endometriosis without endometrioma and 2) deep endometriosis associated with endometriomas.
  * Access to follicular fluid as part of routine care during oocyte retrieval and access to serum as part of routine care during gonadotropin follicular stimulation.
- 4-Infertile Women w/o endometriosis receiving IVF+/-ICSI: Group recruited from the Reproductive Medicine Department : Infertile women without endometriosis receiving IVF+/-ICSI.
  * Women, aged 18-43 receiving IVF± ICSI for female infertility
  * No history of endometriosis or suggestive clinical-biological or radiological signs.
  * The etiology of infertility will be determined in reproductive medicine. Women will be divided into 2 groups of patients:
    1. PCOS (Polycystic Ovary Syndrome). PCOS will be diagnosed in routine care (interrogation, clinical examination, hormone test and pelvic ultrasound) according to the criteria of the Rotterdam Consensus Conference reviewed in 2018.
    2. IOD (Early Ovarian Failure). IOD will be diagnosed in routine care (clinical examination, hormonal and ultrasound check-up) according to the following criteria: AMH<0.8ng/ml and/or CFA <6
  * Access to follicular fluid as part of routine care during oocyte retrieval and access to serum as part of routine care during gonadotropin follicular stimulation
- 5-Fertile W. w/o endometriosis receiving IVF-ICSI as oocyte: Group recruited from the Reproductive Medicine Department : Fertile women without endometriosis receiving IVF-ICSI as oocyte donors.
  * Women receiving IVF± ICSI as oocyte donors
  * No history of endometriosis or clinical-biological or radiological signs suggestive of endometriosis.
  * Access to follicular fluid will be part of the standard care for oocyte puncture and access to serum will be part of the standard care for gonadotropin follicular stimulation.

SUMMARY:
For several years, the effects of environmental pollution on human health have been a growing concern for the scientific community and public authorities. Among the many known chemical contaminants, persistent organic pollutants (POPs) are of particular concern because of their properties as endocrine disrupters, bioaccumulation and biomagnification. The associations between environmental pollutants, endometriosis and infertility remains poorly understood. The objective of this exploratory non interventional monocentric study conducted in the University Hospital of Nantes, is to identify endogenous molecular profiles associated with endometriosis and related infertility. This project implements an exploratory approach combining exposure and metabolomics approaches based on high-resolution mass spectrometry to identify exposure and metabolomics profiles associated with infertility, and biomarkers for potential prognostic application.

DETAILED DESCRIPTION:
LABERCA, a national reference laboratory for chemical pollutants and a labelled metabolomics platform, has developed a new integrative exposure-metabolomics approach based on high-resolution mass spectrometry technologies allowing the exploration of endogenous and exogenous chemical space within biological matrices, coupled with advanced biostatistical methods to promote the identification of biomarkers in health studies (Cano-Sancho et al., 2019). This approach is of great interest both for fundamental research of an etiological and mechanistic nature on complex multifactorial diseases, but also for translational research, which accelerates the application of scientific innovations for better patient care.

Ultimately, the objective is to produce pilot data on the imputability of POPs in infertility and in the pathophysiology of endometriosis in order to reflect on the implementation of preventive measures in infertile women. Identifying exposures to chemical substances and their physiopathological role can help to control their risks and lead to a reflection on the implementation of preventive measures. In case of convincing results, a metabolomic approach will be carried out in order to study the underlying pathogenic mechanisms but also to identify clinical biomarkers. The objective of this project is an integrative multi-omic approach with the ambition to reveal mechanistic associations as well as possible biomarkers of effect on the theme of endometriosis and associated infertility.

This is an observational monocentric non-interventional prospective exploratory study on matched case-control questionnaire and biocollection, in the Reproductive Biology department and in the Gynaecology department of the University Hospital of Nantes.

The biocollection "Obstetrics, Gynaecology and Reproduction", was submitted to the CPP and the CNIL and declared to the Ministry of Research, as well as the informed consent proposed to patients included in our study.

The recruitment of participants is carried out in parallel by the gynaecology department for Groups 1 and 2, and the Reproductive Medicine department for Groups 3, 4 and 5.

The analyses will be carried out by LABERCA. The concentration levels of contaminants will be analyzed by the usual techniques of the LABERCA Laboratory and described in pg or ng per gram of lipid (pg or ng g-1 l w) according to the conventions in force in this field of measurement of lipophilic contaminants, but also in pg or ng per gram of tissue (pg or ng -1 fw) to take into account a mode of expression of the results bearing a complementary level of information The conformity of the analyzed sample and the measurement will be validated by the LABERCA. Measurements of chemical contaminants in the samples from the study will be carried out blindly, and randomly. The analytical methods used by LABERCA to measure the different families of environmental contaminants targeted in this study (historical contaminants such as dioxins, PCBs, PFAS, organochlorine pesticides, or more emerging such as brominated flame retardants, phthalates or bisphenols), are based on high-resolution mass spectrometry-chromatography (GC-HRMS, GC-MS/MS or LC-MS/MS) and isotopic dilution quantification (internal calibration with 13C-labelled compounds), which represents the highest current standard in this field.

The chemical analysis of metabolomic and lipidomic profiles will be performed on the LABERCA metabolomic platform. The platform has developed liquid chromatography methods coupled with high resolution mass spectrometry (LC-HRMS) for non-target profiling from various biological matrices. The analyses will be carried out within an accredited quality management system (ISO 9001 and IBISA)

ELIGIBILITY:
Inclusion Criteria :

* Women aged 18 to 45 years benefiting from surgery in the Gynaecology-Obstetrics department or IVF± ICSI (In Vitro Fertilization+/- Intracytoplasmic Injection of Spermatozoid) in the Medicine and Reproductive Biology department of the University Hospital of Nantes.
* No objection to participate in the study
* Collection of consent for the Gynaecology-Obstetrics Bio-collection

Group 1 - Women without deep endometriosis benefiting surgery :

* Caucasian women, aged 18 to 45 years undergoing gynaecological surgery, for example: benign laparoscopy (example: tubal ligation), benign ovarian surgeries or benign uterine procedures (fibroma, ovarian cyst) or genital prolapse.
* Non-interventional access to parietal and epiploic adipose tissue as part of routine care
* No clinical-biological criteria in favour of a diagnosis of endometriotic disease, nor any radiological evidence (ultrasound or MRI) suggestive of endometriosis.

Group 2 - Women with endometriosis benefiting surgery :

* Caucasian women aged 18 to 45
* Severe and deep endometriotic pathology, with or without endometriomas, with surgical indication (clinical examination, imaging examinations, intraoperative observation),
* Access to epiploid and/or parietal adipose tissue as part of routine care.

Group 3 - Infertile women with deep endometriosis benefiting from IVF :

* Women with IVF or ICSI for infertility with deep endometriosis diagnosed in routine care (clinical examination, imaging examinations +/- surgical findings). They will be classified into 2 subgroups: 1) deep endometriosis without endometrioma and 2) deep endometriosis associated with endometriomas.
* Access to follicular fluid as part of routine care during oocyte retrieval and access to serum as part of routine care during gonadotropin follicular stimulation.

Group 4 - Infertile women without endometriosis receiving IVF+/-ICSI :

* Women, aged 18-43 receiving IVF± ICSI for female infertility
* No history of endometriosis or suggestive clinical-biological or radiological signs.
* The etiology of infertility will be determined in reproductive medicine. Women will be divided into 2 groups of patients :

  1. PCOS (Polycystic Ovary Syndrome). PCOS will be diagnosed in routine care (interrogation, clinical examination, hormone test and pelvic ultrasound) according to the criteria of the Rotterdam Consensus Conference reviewed in 2018.
  2. IOD (Early Ovarian Failure). IOD will be diagnosed in routine care (clinical examination, hormonal and ultrasound check-up) according to the following criteria: AMH<0.8ng/ml and/or CFA <6
* Access to follicular fluid as part of routine care during oocyte retrieval and access to serum as part of routine care during gonadotropin follicular stimulation

Group 5 - Fertile women without endometriosis receiving IVF-ICSI as oocyte donors :

* Women receiving IVF± ICSI as oocyte donors
* No history of endometriosis or clinical-biological or radiological signs suggestive of endometriosis.
* Access to follicular fluid will be part of the standard care for oocyte puncture and access to serum will be part of the standard care for gonadotropin follicular stimulation.

Cases' exclusion criteria :

* Opposition from the patient.
* Intercurrent diagnosis of pregnancy incompatible with surgery or IVF+/-ICSI

Controls ' exclusion criteria :

* Clinical or radiological signs suggestive of endometriosis
* Opposition from the patient.
* Intercurrent diagnosis of pregnancy incompatible with surgery or IVF+/-ICSI

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Women recruited in the Gynaecology-Obstetrics and Reproductive Medicine Departments
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Identify endogenous molecular profiles of patients with infertile endometriosis | baseline
  Statistical associations between exposomics and presence of deep endometriosis with infertility

SECONDARY OUTCOMES:
Characterize the internal chemical exposure profiles and metabolomic profiles in the different groups. | baseline
  Statistical differences between exposome and metabolome molecular signatures between subgroups of the study populations.
Compare the distribution of contaminant concentration levels and metabolomic profiles according to the media measured. | baseline
  Statistical correlations between exposome and metabolome molecular signatures between sampling sites

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No